CLINICAL TRIAL: NCT01793662
Title: Norwegian Laparoscopic Aortic Surgery Trial
Acronym: NLAST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Syed Sajid Hussain Kazmi, Consultant Surgeon, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NLAST2012
Record Dates: First submitted 2013-02-14; First posted 2013-02-15 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Aortobifemoral Bypass; Aortoiliac Occlusive Disease; TASC Type D Lesions; Laparoscopic Versus Open Bifurcation Graft
Keywords: Aortobifemoral bypass; Laparoscopic aortic surgery; Aortoiliac occlusive disease; TASC Type D Lesions; Open aortic surgery
MeSH Terms: interventions — Laparoscopes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Open aortobifemoral bypass (Active Comparator): Patients with aortoiliac occlusive disease (only, TASC Type D lesions) shall be randomized to either laparoscopic aortobifemoral bypass or open aortobifemoral bypass operation.
  Interventions: Procedure: Laparoscopic aortobifemoral bypass
- Laparoscopic aortobifemoral bypass (Experimental): Patients with aortoiliac occlusive disease (only, TASC Type D lesions) shall be randomized to either laparoscopic aortobifemoral bypass or open aortobifemoral bypass operation.
  Interventions: Procedure: Laparoscopic aortobifemoral bypass

INTERVENTIONS:
Procedure: Laparoscopic aortobifemoral bypass — Totally laparoscopic aortobifemoral bypass shall be performed and the patients in this intervention arm shall be compared with the control arm randomized for open aortobifemoral bypass operation.
  Other Names: Laparoscopic aortic surgery; laparoscope

SUMMARY:
Patients with severe atherosclerotic occlusive disease can be operated on with an aortobifemoral bypass(ABFB)through a median laparotomy. Since 1993, this operation has also been performed laparoscopically. The laparoscopic ABFB operation claims to be minimally invasive as compared to the open ABFB. The cohort studies published so far have shown that although a longer operation time with the laparoscopic procedure as compared to the open surgery, the patients have a shorter hospital stay, lesser perioperative bleeding, fewer systemic complications, and earlier convalescence.

However, no randomized control trial has yet been published to compare the two procedures.

In the NLAST-study, which is a multicenter randomized control trial, the patients with TASC type D atherosclerotic lesions shall be randomized to either totally laparoscopic aortobifemoral bypass operation (LABFB)or an open ABFB operation.

DETAILED DESCRIPTION:
The primary endpoint of the study is post-operative complications defined as systemic and local complications, including vascular complications e.g., graft infection, thrombosis, etc.

Secondary endpoints are as follows,

* health-related quality of life, examined and evaluated with the help of pre and post-operative surveys performed with the help of SF36v2 questionnaire and EQ5D5L.
* perioperative stress response (during operation) measured/analyzed with the help of stress hormones changes
* perioperative inflammatory response
* cost-utility analysis
* cost differences

ELIGIBILITY:
Inclusion Criteria:

* Aortoiliac occlusive disease (TASC Type D lesions)

Exclusion Criteria:

* Active cancer disease
* Acute critical limb ischemia
* Prior major abdominal surgery
* Heart failure (Ejection fraction <40%

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2013-02; Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | 2.9 years
  Postoperative complications during a mean follow-up period of 2.9 years are the primary outcome measure of NLAST.

SECONDARY OUTCOMES:
health related quality of life | 3 months postoperatively
  The bodily pain domain of the SF36-v2 at 3 months postoperatively shall be used to assess the patients in the two groups of NLAST study. Besides EQ-5D-5L shall be used pre and post operatively for QoL evaluation.

OTHER OUTCOMES:
Operative stress response | During operation
  During operation changes in the stress hormones e.g., adrenalin, cortisol etc shall be analyzed in the two patients groups.
Cost utility examination | 30 days
  In hospital cost of the treatment shall be calculated. Cost utility examination shall be performed.
Inflammatory stress response | 30 days
  Changes in the pro-inflammatory interleukins etc shall be registered during and after operation.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Sajid Hussain Kazmi, MD, PhD, Principal Investigator — Department of vascular surgery, Oslo University Hospital, Oslo, Norway
Locations (1):
- Department of vascular surgery, Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kazmi SSH, Sahba M, Pettersen EM, Krog AH, Fagerland MW, Sundhagen JO. Norwegian Randomised Trial of Laparoscopic versus Open Aortobifemoral Bypass: The Norwegian Laparoscopic Aortic Surgery Trial (NLAST). Eur J Vasc Endovasc Surg. 2025 Nov 7:S1078-5884(25)00932-3. doi: 10.1016/j.ejvs.2025.09.046. Online ahead of print. PMID 41207501

DOCUMENTS (2):
  • Study Protocol (2013-02-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT01793662/Prot_001.pdf
  • Statistical Analysis Plan (2025-06-26): https://cdn.clinicaltrials.gov/large-docs/62/NCT01793662/SAP_002.pdf